CLINICAL TRIAL: NCT06261398
Title: Better Birth Outcomes and Experiences Through Technology, Education, and Reporting (BETTER)
Brief Title: Better Birth Outcomes Through Technology, Education, and Reporting
Acronym: BETTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Ann McAlearney, Professor of Family Medicine and Executive Director, CATALYST, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023H0065
Record Dates: First submitted 2024-01-31; First posted 2024-02-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy; Maternal Anemia; Pre-Term Birth; Hypertensive Disorders
Keywords: Social Determinants of Health (SDoH); Pregnancy; Patient portals; Patient engagement; Disparities
MeSH Terms: conditions — Patient Participation | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BETTER Intervention (Experimental): Patients in the intervention group will receive one motivational interviewing session immediately after randomization and biweekly text messages until delivery to encourage them to connect to resources to address their social needs.
  Interventions: Behavioral: BETTER: motivational interviewing and text messaging
- Standard of care (Active Comparator): No motivational interviewing or text messages will be provided.
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: BETTER: motivational interviewing and text messaging — Motivational interviewing to encourage individuals to address their social needs and engage with text messages that allow individuals to connect to their care team, a local organization that can help them address their social needs, and/or a resource that enables them to find help to address their needs based on their zip code.
  Arms: BETTER Intervention
Behavioral: Standard of care — No motivational interviewing or text messages will be provided.
  Arms: Standard of care

SUMMARY:
This is a pragmatic randomized control trial to evaluate the BETTER intervention compared to standard obstetrical care (control) to determine whether it helps to reduce maternal anemia and other adverse pregnancy outcomes. The BETTER intervention includes one motivational interviewing session and bi-weekly text messages to encourage patients to connect with resources that address their social needs, including housing, food, and transportation. Quantitative data will be used to study participant outcomes, including surveys, and electronic health record data.

DETAILED DESCRIPTION:
There are more than 3.5 million births per year in the United States. A substantial portion of these births (approximately 25-30%) occur in the context of significant adverse pregnancy outcomes (APOs) including preterm birth (PTB), hypertensive disorders of pregnancy (HDP), small-for-gestational-age birth (SGA), and intrauterine fetal demise (IUFD). Moreover, these complications significantly increase the risk of both maternal and perinatal morbidity and mortality and are associated with adverse health consequences throughout the life course of both individuals. Anemia in pregnancy has been consistently cited as an important factor in and upstream of APOs such as PTB and HDP, severe maternal morbidity, and maternal mortality, and for disparities in these outcomes as well.

This study will expand our understanding of addressing SDoH, including linkage to services that mitigate SDoH. This information can inform future interventions that address SDoH. Creating new tools to address the needs and strengths of obstetric patients, and encouraging their use, will improve the management of patient care during and after pregnancy.

The patient sample will include obstetric patients receiving care at the OSUWMC McCampbell OB/GYN clinic or the OSUWMC Outpatient Care East OB/GYN clinic. A total of 550 patients will participate in the study and be randomly assigned to either the intervention or control group. We will collect maternal and child health outcome data using patient electronic health records and surveys.

At the time of randomization at the patient's prenatal appointment, a researcher will use a survey to collect participant baseline data, including patient demographics and patient-reported outcomes. This information will be collected again during a study visit during the patient's prenatal appointment when the patient is 28-32 weeks gestation.

Final data collection from patient records will occur after delivery (for both intervention and control groups). Research staff will extract information from patients' and their baby's medical records, including maternal and perinatal outcomes.

The intervention includes one motivational interviewing session that encourages the patient to address their social needs. Following the intervention, patients will receive bi-weekly text messages with links to help them address social needs; these links are: (1) to a patient portal to enable them connect with their care team, (2) to Health Impact Ohio, a local organization that can help patients address social needs; and (3) to "findhelp.org," a site that can provide a list of resources based on zip code.

ELIGIBILITY:
Inclusion Criteria

* Less than 20 weeks and 6 days pregnant upon enrollment
* At least 18 years of age
* Receiving obstetric care at OSU McCampbell Hall or OSU Outpatient Care East
* Singleton pregnancy and fetus with a heartbeat
* English speaking
* Able to receive text messages

Exclusion Criteria

* Has a significant medical condition (eg sickle cell disease) that is a cause of anemia
* Has a plan for transfusion during pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is restricted to pregnant individuals.
Enrollment: 550 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of maternal anemia | At delivery
  Hemoglobin < 11.0 g/dL

SECONDARY OUTCOMES:
Incidence of Pre-term birth | At delivery
  Delivery prior to 37 weeks of gestation
Incidence of Hypertensive disorders of pregnancy | Through study completion, approximately 6 months
  Antepartum gestational hypertension or preeclampsia of any severity through the postpartum
Incidence of infection | Through study completion, approximately 6 months
  As determined by clinical diagnosis (e.g., chorioamnionitis, endometritis, pyelonephritis); intrapartum and postpartum
Incidence of Cesarean Delivery | At delivery
  Delivery by Cesarean section
Incidence of Postpartum hemorrhage | Through study completion, approximately 6 months
  Blood loss >1000cc
Incidence Severe maternal morbidity | Through study completion, approximately 6 months
  >3 units of packed red blood cell transfusion or ICU admission
Incidence of maternal mortality | Through study completion, approximately 6 months
  Death
Incidence of Small for gestational age birth | At birth
  <10th percentile for gestational age
Incidence of Large for gestational age | At birth
  >90th percentile for gestational age
Incidence of NICU admission | Through study completion, approximately 6 months
  Admission to the NICU
Incidence of Perinatal mortality | Through study completion, approximately 6 months
  Intrauterine or neonatal death
Incidence of Prenatal care visits | From randomization through delivery
  Number of prenatal care visits
Incidence of Antepartum admission | From randomization through delivery
  Hospital admission other than for delivery
Length of stay (days) | Immediately after discharge from the delivery hospitalization
  Length of hospital stay at delivery admission
Postpartum re-admission | From delivery discharge through 6 weeks post partum
  Hospital admission after postpartum discharge

CONTACTS AND LOCATIONS:
Overall Officials: William Grobman, MD, MBA, Principal Investigator — Ohio State University; Ann McAlearney, ScD, MS, Principal Investigator — Ohio State University
Locations (3):
- United States (3):
  - The Ohio State University Outpatient Care East, Columbus, Ohio
  - McCampbell Hall, Columbus, Ohio
  - The Ohio State University Wexner Medical Center OB/GYN Maternal and Fetal Medicine, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McAlearney AS, MacEwan SR, Huerta TR, Thomas NR, Sova LN, Roth L, Bartholomew A, Rush LJ, Johnson KF, Grobman WA. Patient-informed outpatient intervention to improve pregnancy outcomes through connections to social services: protocol for the BETTER randomised controlled trial. BMJ Open. 2025 Jun 18;15(6):e096119. doi: 10.1136/bmjopen-2024-096119. PMID 40533225